## A Home-based Video and Motivational Interviewing Intervention to Improve Preschoolers Diet Quality and Parental Food Parenting Practices Statistical Analysis Plan

NCT03923491

ID: 1R34HL140229-01A1

Date of Analysis Plan: May 18, 2020

We will assess for between-group differences in baseline characteristics (demographics) using graphical methods, non- parametric and parametric tests as appropriate (e.g., Wilcox in rank-sum test for skewed data, t-tests for normally distributed continuous data and chi-squared tests for categorical data) and variables found to be important covariates will be included in subsequent analyses. We will estimate the preliminary efficacy of the intervention compared to comparison using a generalized linear model in which we will compare 6-month HEI, feeding and food availability between study conditions, while controlling for baseline HEI, feeding and food availability scores and potential confounders. Modeling will be done using a likelihood-based approach and thus makes use of all available data. Inverse Probability of Retention Weighting (IPRW) will be used to reduce selection bias due to non-response. In addition, any variables with persistent imbalances between responders and non-responders after IPRW will be added to each outcome model to help control for any residual bias due to selective attrition. We are aware that effect size estimates with small samples have large standard errors and wide confidence intervals and expect this to be the case in this pilot trail.